CLINICAL TRIAL: NCT06757062
Title: Less Pain, More Game: Efficacy of Red Kinesiology Tape on Carpal Tunnel-Like Symptoms and Performance in Esports Gamers
Brief Title: Efficacy of Red Kinesiology Tape on Carpal Tunnel-Like Symptoms and Performance in Esports Gamers
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nevada, Las Vegas (Other)
Responsible Party: Principal Investigator, Donnamarie Krause, PhD, OTR/L, Director Doctor of Occupational Therapy Programs, Principal Investigator, Associate Professor, University of Nevada, Las Vegas
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: UNLV-2024-431
Record Dates: First submitted 2024-12-09; First posted 2025-01-03 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Carpal Tunnel Syndrome
Keywords: Esports; Gamers; Carapl Tunnel Syndrome; Performance; First Person Shooter; Red; Color Theory; Kinesio Tape; Kinesiology Tape; Dorsal Application
MeSH Terms: conditions — Carpal Tunnel Syndrome; Erythema

STUDY DESIGN:
Intervention Model Description: Participation in this study requires 2 visits to the UNLV Shadow Lane Campus OT Skills Lab located at 1125 Shadow Ln, Las Vegas, NV 89102. Visits will require no more than 60 minutes of the participant's time and involve kinesiology tape applications, quick performance measures, and questionnaires.
  This study follows a randomized controlled crossover design with 2 study arms: red KT and skin tone KT. Each intervention will be applied once and separated by a washout period which will be at least 1 week.
  Participants will be randomly assigned to either group X or group Y, indicating their sequence of receiving the two treatments. Group X would receive red KT then skin tone KT while group Y would receive skin tone KT then red KT. This will be done by having the participant select an envelope containing one of the two group assignments.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Red Kinesiology Tape Applied with the Dorsal Application for Carpal Tunnel Syndrome (Experimental): The red kinesiology tape will be applied with the dorsal application for carpal tunnel syndrome. It is explained and utilized in Krause et al. (2020). The color red has been found in previous studies to impact motor function and performance in various activities specifically when looking at activities of an aggressive or competitive nature. Thus red was chosen when assessing the color effect of red in first-person shooter games which require outperforming the opponent with quick reaction time, accuracy, and aggression.
  Each participant will receive the red KT application only once. The order of which they receive the red KT or the skin tone KT will depend on their random assignment to group X or Y.
  The KT will be applied by an interventionist trained in proper KT application. Participants will be educated on self-removal specifically given by the manufacturer of the brand of KT used (Sparthos Tape). There will be a 7 day washout period between tape applications.
  Interventions: Device: Kinesiology Tape
- Skin Tone Kinesiology Tape Applied with the Dorsal Application for Carpal Tunnel Syndrome (Active Comparator): The skin tone kinesiology tape will be applied with the dorsal application for carpal tunnel syndrome. It is explained and utilized in Krause et al. (2020). Sparthos KT offers skin tone KT covering multiple shades to allow the closest color to match the participant's skin. Utilizing other skin tones other than beige allows inclusion and diversity. The skin tone KT was chosen to diminish the effect of the KT color to allow better isolation and study of the effect of the color red in comparison.
  Each participant will receive the skin tone KT application only once. The order in which they receive the red KT or the skin tone KT will depend on their random assignment to group X or Y.
  The KT will be applied by an interventionist trained in proper KT application. Participants will be educated on self-removal specifically given by the manufacturer of the brand of KT used (Sparthos Tape). There will be a 7 day washout period between tape applications.
  Interventions: Device: Kinesiology Tape

INTERVENTIONS:
Device: Kinesiology Tape — The kinesiology tape (KT) is applied with the dorsal application for the treatment of carpal tunnel syndrome (CTS). This method is utilized and explained in Krause et al. (2020). This study will assess the efficacy of the application method as well as the varying effects of the color of the KT. Red KT will be compared to skin tone KT. The skin tone KT will be color-matched as closely as possible to each participant's skin tone to reduce the effect of the KT color. In this way, the study's second purpose is to understand the potential effect of color on psychological function and performance in the context of aggressive first-person shooter esports games.

SUMMARY:
The goal of this clinical trial is to learn if dorsally applied kinesiology tape is an effective conservative treatment for symptoms of carpal tunnel syndrome and assess the potential performance effect of the tape color in first-person shooter esports games in esports gamers who exhibit symptoms that resemble carpal tunnel syndrome. The main questions it aims to answer are:

Is dorsally applied kinesiology tape able to manage carpal tunnel syndrome-like symptoms in esports gamers? Does red kinesiology tape hinder or improve performance in first-person shooter esports games in esports gamers?

Researchers will compare red kinesiology tape to skin tone kinesiology tape. Both will be applied on the dorsal aspect of the hand and wrist of the dominant upper extremity.

Participants will visit the site 2 times to get kinesiology tape applied and complete a pre and post-test for pain and performance. Depending on randomization a participant will receive a random sequence of the study arm (ex: red then skin tone or skin tone then red tape)

DETAILED DESCRIPTION:
Less Pain, More Game - Efficacy of Red Kinesiology Tape on Carpal Tunnel Symptoms and Performance in Esports Gamers is a clinical trial that aims to determine if dorsally applied kinesiology tape can manage or improve symptoms that resemble carpal tunnel syndrome in esports gamers. Esports gamers use their hands very differently from the average individual when participating in hours of video game play. This study first aims to test if kinesiology tape would benefit these individuals despite the frequency and intensity with which they use their hands and fingers.

Performance and competition is a major component of esports gaming participation. Despite how well kinesiology tape may improve symptoms of carpal tunnel syndrome, it would not be a good treatment option if it hindered their ability to participate in esports. This study also aims to address performance as well. Color has been identified as a quality of kinesiology tape that may impact performance. Thus this study also seeks to assess the potential performance effect of the tape color in first-person shooter esports games in esports gamers who exhibit symptoms that resemble carpal tunnel syndrome.

Participants will visit the site 2 times to get kinesiology tape applied and complete a pre and post-test for the Short Form Mcgill Pain Questionnaire and a first-person shooter simulation to assess performance. The study design is a randomized controlled crossover trial thus depending on randomization a participant will receive a random sequence of the study arm (ex: red then skin tone or skin tone then red tape).

Results from this study would allow occupational therapists to promote health and wellness within the esports gamer population and enhance performance to give players an edge over their opponents.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years old
* can see color vision
* reports having numbness, tingling, weakness, or pain in the hands, wrist, or fingers
* has a positive Phalen's test result
* passes Ishihara Color Vision Test with a score of at least 12
* provides written consent
* reports to play video games over 5 hours a week on average

Exclusion Criteria:

* cognitively impaired
* pregnant
* has history of skin conditions
* has history of hand conditions other than carpal tunnel syndrome
* has history of surgery to the wrist, hand, or fingers
* is currently receiving other forms of physiotherapy
* has open wounds on the kinesiology tape application site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-01-01 (Estimated); Primary Completion 2025-03-30 (Estimated); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
McGill Pain Questionnaire Short-Form | at intervals throughout the 3 week cycle
  Short Form - McGill Pain Questionnaire - 2 will give outcomes of pain intensity and quality. It includes adjectives to describe both nociceptive pain and neuropathic pain. Pain descriptors can be categorized into Continuous (throbbing pain, cramping pain, gnawing pain, aching pain, heavy pain, tender), Intermittent (shooting pain, stabbing pain, sharp pain, splitting pain, electric-shock pain, piercing), Neuropathic (hot-burning pain, cold-freezing pain, pain caused by light touch, itching, tingling or "pins and needles", numbness), and Affective (tiring-exhausting, sickening, fearful, punishing-cruel)
  It will be taken 4 times by each participant: before the first application of the KT, after the first application of the KT, before the second application of the KT in the opposite color, and after the second application of the KT in the opposite color.

SECONDARY OUTCOMES:
3D Aim Trainer Attack Bombsite Simulation | at intervals throughout the 3 week cycle
  It is an esports shooting simulation on easy difficulty and is completed on a Dell PC with a keyboard and mouse setup. It will measure performance through a collection of overall scores and accuracy percentages. The participants will have to shoot at enemy targets while dodging attacks and surviving to the next stage. Each stage of the simulation will increase in difficulty. The simulation will be completed with the computer set to a grayscale display to eliminate any effect of the colors of the original simulation. Each attempt of the simulation will end after 200 seconds. It will be completed in a private room with only the student researcher present. The simulation is free and can be found here: https://www.3daimtrainer.com/. Data from this simulation will be stored under the participant ID code on a protected Google Sheets document.
  It will be taken 4 times by each participant: before KT, after the KT, before the KT in the opposite color, and after KT in the opposite color.

OTHER OUTCOMES:
End of Study Survey | at the last visit of the 3-week study cycle
  It is completed only once online after self-removal of the 2nd KT application. This survey will ask about how long the tape lasted before it lost adhesiveness, KT color preference, willingness to recommend KT to others, KT color effect on performance, and KT color effect on CTS symptoms. This will be completed anonymously on their own time as an additional component of the study to collect qualitative comments related to their experience with the KT. They will also be able to indicate their desire to learn how to self-apply KT. If they indicate an interest in self-application, they will be directed to email the student researcher.

CONTACTS AND LOCATIONS:
Overall Officials: Donnamarie Krause, Ph.D, Principal Investigator — University of Nevada, Las Vegas
Locations (1):
- University of Nevada, Las Vegas - Shadow Lane Campus, Las Vegas, Nevada, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Krause D, Roll SC, Javaherian-Dysinger H, Daher N. Comparative efficacy of the dorsal application of Kinesio tape and splinting for carpal tunnel syndrome: A randomized controlled trial. J Hand Ther. 2021 Jul-Sep;34(3):351-361. doi: 10.1016/j.jht.2020.03.010. Epub 2020 Sep 4. PMID 32893100

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2024-11-14): https://cdn.clinicaltrials.gov/large-docs/62/NCT06757062/Prot_SAP_ICF_000.pdf